CLINICAL TRIAL: NCT05962593
Title: Surgical Removal of Mandibular Third Molars. Inflammation, Infection, Pain and Complications. Different Inflammatory Biomarkers With Surgical Removal of Mandibular Third Molars
Brief Title: Different Inflammatory Biomarkers With Surgical Removal of Mandibular Third Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H 22029533
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Wisdom Teeth
Keywords: wisdom teeth; inflamation; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telephone call (Placebo Comparator): A postoperative telephone call
  Interventions: Other: Telephone call
- No telephone call (No Intervention): No telephone call

INTERVENTIONS:
Other: Telephone call — The patients will be randomized for a postoperative telephone call
  Arms: Telephone call

SUMMARY:
Removal of mandibular third molars (M3s) is the most frequently performed surgical intervention undertaken in dentistry. The indications and timing of surgical removal of M3s has been a matter of international and national debate, and especially prophylactic removal of M3s is controversial.

DETAILED DESCRIPTION:
Removal of mandibular third molars (M3s) is the most frequently performed surgical intervention undertaken in dentistry. The indications and timing of surgical removal of M3s has been a matter of international and national debate, and especially prophylactic removal of M3s is controversial.

It is well documented that periodontally compromised patients are characterized by elevated levels of systemic low-grade inflammation which can affect their general health and contribute to development and aggravation of a number of chronic diseases including diabetes mellitus and cardiovascular disorders. Inflammatory changes are frequent around erupted, semi-erupted and retained M3s. However, only a few under-powered studies have addressed the relationship between the presence of M3s and the level of systemic low-grade inflammation.

Conservative guidelines recommend not to remove M3s until subjective and/or objective signs of infection are observed. Overall, these guidelines result in a relatively equal distribution of surgically removed M3s over the age span of a population. In contrast, more proactive guidelines recommend removal of M3s that are not expected to erupt into functional occlusion leading to frequent removal of M3s in the young population. Surgical removal of M3s are associated with a varying degree of pain, facial swelling and the patients are on average sick leave for 2-3 days. Furthermore, complications as nerve damage, infection, bleeding and jaw fracture can occur. Therefore, unnecessary removal of M3s should be avoided. However, the risk and severity of postoperative sequelae and complications is known to increase significantly with age. Hence, the crucial point determining indications for surgical removal of M3s is to balance the risk of developing local and systemic disease against the risk of complications after surgical removal.

The present project will investigate the systemic impact of retaining or removing M3s by measuring low-grade systemic inflammation markers in blood and saliva. To further explore measures to reduce postoperative complications, discomfort, and patient satisfaction, the effect of prophylactic antibiotics, pre-emptive analgesics, and a postoperative follow-up telephone call, will be investigated.

The project consists of six prospective studies that will include more than 800 patients and surgical removal of more than 1,000 mandibular third molars. It is expected that the project will contribute with important information on the impact of mandibular third molars on general health and prophylactic modalities that can influence postoperative sequelae and complications following surgical removal of mandibular third molars.

ELIGIBILITY:
Inclusion Criteria:

* Wisdom teeth

Exclusion Criteria:

* No wisdom teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Inflammation | 3 months postoperative
  High sensitive C-reactive protein

SECONDARY OUTCOMES:
Pain score | 1-7 days postoperative
  NRS

CONTACTS AND LOCATIONS:
Overall Officials: Marie Kj Larsen, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark